CLINICAL TRIAL: NCT02224521
Title: An Open-label, Randomised, Single-dose, Multi-cohort, Crossover Bioavailability Study of a Solution Formulation and Three Capsule Formulations of GSK2190915 in Healthy Adult Subjects Followed by a Repeat-dose, Randomized, Parallel Group, Double-blinded Study of One Selected Capsule Formulation and Matched Placebo in Elderly Healthy Subjects
Brief Title: GSK2190915A - Bioavailability Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 112071
Record Dates: First submitted 2011-06-23; First posted 2014-08-25 (Estimated); Last update posted 2017-06-14 (Actual); Status verified 2017-06

CONDITIONS: Asthma
Keywords: FLAP inhibitor; Chronic Obstructive Pulmonary Disease (COPD); COPD; Bioavailability
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Cohort 1 (Experimental): Subjects will be assigned to any of the 4 dosage regimen (A, B, C, D) in four periods. A= GSK2190915 Solution, 50mg single dose, fasted; B = GSK2190915 Capsule Formulation A, 50mg single dose (1 x 50mg capsule), fasted; C= GSK2190915 Capsule Formulation B, 50mg single dose (1 x 50mg capsule), fasted; D= GSK2190915 Capsule Formulation C, 50mg single dose (1 x 50mg capsule), fasted.
  Interventions: Drug: GSK2190915 Solution.; Drug: GSK2190915 Granule Capsule (A); Drug: GSK2190915 Semi-solid Lipid Capsule (B); Drug: GSK2190915 Liquid Lipid Capsule (C)
- Cohort 2 (Experimental): The selected formulation will be dosed with GSK2190915 capsule formulation at 20mg (fasted), 100mg (fasted), 100mg (fed) and 200mg (fasted).
  Interventions: Drug: GSK2190915 Solution.; Drug: GSK2190915 Granule Capsule (A); Drug: GSK2190915 Semi-solid Lipid Capsule (B); Drug: GSK2190915 Liquid Lipid Capsule (C)
- Cohort 3 (Experimental): Cohort 3 will be a 4-way complete crossover study with single doses of 20mg and 200mg of up to two capsule formulations taken forward from cohort 2 in 10 healthy adult subjects in the fasted state.
  Interventions: Drug: GSK2190915 Solution.; Drug: GSK2190915 Granule Capsule (A); Drug: GSK2190915 Semi-solid Lipid Capsule (B); Drug: GSK2190915 Liquid Lipid Capsule (C)
- Cohort 4 (Experimental): The regimen for Cohort 4 will be either the highest dose (200mg) of the capsule formulation (A, B or C) taken forward from the previous cohorts or the solution formulation (200mg).
  Interventions: Drug: GSK2190915 Solution.; Drug: GSK2190915 Granule Capsule (A); Drug: GSK2190915 Semi-solid Lipid Capsule (B); Drug: GSK2190915 Liquid Lipid Capsule (C)
- Cohort 5 (Experimental): Subjects will take milled and micronised tablet formulations of GSK2190915 in the fasted state in periods 1 and 2, and will take milled and micronised tablet formulations of GS2190915 in the fed state in periods 3 and 4.
  Interventions: Drug: GSK2190915 Milled Tablet; Drug: GSK2190915 Micronised Tablet
- Cohort 6 (Experimental): Tablet formulations (milled and micronised, different to the Cohort 5 formulations) of GSK2190915 will be dosed in the fasted and fed (after a light breakfast) states.
  Interventions: Drug: GSK2190915 Milled Tablet; Drug: GSK2190915 Micronised Tablet

INTERVENTIONS:
Drug: GSK2190915 Solution. — Aqueous Solution, 10mg/mL.
  Arms: Cohort 1; Cohort 2; Cohort 3; Cohort 4
Drug: GSK2190915 Granule Capsule (A) — GSK2190915A granule filled in to Gelatin capsules
  Arms: Cohort 1; Cohort 2; Cohort 3; Cohort 4
Drug: GSK2190915 Semi-solid Lipid Capsule (B) — GSK2190915A dispersed in a lipid vehicle and filled in to HPMC capsules
  Arms: Cohort 1; Cohort 2; Cohort 3; Cohort 4
Drug: GSK2190915 Liquid Lipid Capsule (C) — GSK2190915A dissolved in lipid vehicle milled and filled in to Gelatin capsules
  Arms: Cohort 1; Cohort 2; Cohort 3; Cohort 4
Drug: GSK2190915 Milled Tablet — GSK2190915A granule is blended, compressed into tablets and aqueous film coated
  Arms: Cohort 5; Cohort 6
Drug: GSK2190915 Micronised Tablet — GSK2190915A granule is blended, compressed into tablets and aqueous film coated
  Arms: Cohort 5; Cohort 6

SUMMARY:
GSK2190915 is a high affinity 5-lipoxygenase-activating protein (FLAP) inhibitor that reduces inflammation in cells.

This study will evaluate three capsule and two tablet formulations to select the optimal formulation for further development. Safety will be assessed through clinical laboratory testing, 12-lead electrocardiogram (ECG), vital signs and Adverse Event/ Serious Adverse Event (AE/ SAE) recording.

DETAILED DESCRIPTION:
GSK2190915 is a high affinity 5-lipoxygenase-activating protein (FLAP) inhibitor that attenuates the production of leukotrienes, through the blockage of the first committed step in the leukotriene pathway, 5 lipoxygenase (5-LO) activation. Leukotrienes are potent inflammatory molecules produced mainly by mast cells, eosinophils, monocytes/macrophage and neutrophils in response to allergic or inflammatory stimuli.

Clinical studies conducted to date with GSK2190915 have utilised an aqueous formulation of the compound. However, to progress the compound further in clinical development, a solid dose formulation is necessary. This study will evaluate the optimal capsule formulation from a selection of three available capsule formulations, and a dose, that can be taken forward for future clinical development. Since it is expected that the compound will be developed for Chronic Obstructive Pulmonary Disease (COPD), the study will also include a repeat-dose cohort with elderly subjects (smokers and non-smokers over 65 years of age) in order to evaluate the repeat-dose derived pharmacokinetic parameters of the selected capsule formulation in this population.

This is a multi-cohort study and upto 6 cohorts will be performed.

In cohort 1, the bioavailability of single doses of 50 milligrammes (50 mg) of three capsule formulations (capsule formulations A, B and C) in the fasted state will be assessed. Depending on the bioavailability data obtained from cohort 1, one, two or three capsule formulations may be taken forward into cohort 2.

If only one formulation is deemed to be suitable for progression, cohort 2 will be a single-dose, 4-way complete crossover study to investigate both food-effect and dose proportionality in 10 healthy adult subjects. The decision to progress this formulation to the final (repeat-dose) cohort (cohort 4) will be made based on favourable food interaction and proportionality in bioavailability between high and low doses in cohort 2.

If more than one capsule formulation fulfils the bioavailability criteria following cohort 1, cohort 2 will be a food-effect study with a 100mg single dose of two or three selected capsule formulations in healthy adult subjects. Progression to Cohort 3 will be dependent on the formulation/s meeting predetermined pharmacokinetic (PK) criteria. Cohort 3 will be a complete crossover study with single doses of 20mg and 200mg of each of upto two capsule formulations taken forward from cohort 2 in 10 healthy adult subjects in the fasted state. The aim of performing this cohort is to explore the dose proportionality between low and high doses of the two selected capsule formulations.

Cohort 4 is a 12-day repeat-dose, double-blinded, placebo-controlled study in 12 healthy elderly subjects (>65 years) in the fed or fasted state with once-daily dosing of the highest dose (200mg) of the capsule formulation (A, B or C) taken forward from the previous cohorts. The aim of this cohort is to investigate the accumulation of the selected formulation during repeat dosing.

Cohort 5 will be a 4-way complete crossover study with single doses of 100mg of two tablet formulations (milled and micronised) administered to healthy volunteers in the fed and fasted states. The aim of performing this cohort is to explore the single-dose pharmacokinetics of the two tablet formulations with a view to assessing their suitability for use in subsequent late- phase studies.

Cohort 6 will be a 4-way complete crossover study with single doses of 100mg of two modified tablet formulations (different from Cohort 5 formulations) administered to healthy volunteers in the fed and fasted states. The aim of performing this cohort is to explore the single-dose pharmacokinetics of the two modified tablet formulations with a view to assessing their suitability for use in subsequent late- phase studies.

ELIGIBILITY:
Inclusion Criteria:

INCLUSION CRITERIA FOR COHORTS 1, 2, 3, 5 and 6.

A subject will be eligible for inclusion in cohorts 1, 2, 3, 5 and 6 of this study only if all of the following criteria apply:

1. Aspartate transaminase (AST), alanine transaminase (ALT), alkaline phosphatase and bilirubin less than or equal to 1.5 times Upper Limit of Normal, ULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin less than 35 percent).
2. Healthy as determined by the Investigator, based on a medical evaluation including medical history, physical examination, laboratory tests and Electrocardiogram (ECG). A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included only if the Investigator and the GSK Medical Monitor agree that the finding is unlikely to introduce additional risk factors and will not interfere with the study objectives.
3. Male or female (of non child-bearing potential) between 18 and 65 years of age inclusive, at the time of signing the informed consent.

   A female subject is eligible to participate only if she is of:

   •Non-childbearing potential defined as pre-menopausal females with a documented tubal ligation (in which case the male partner should use an acceptable form of contraception as specified in section 8.1) or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) > 40 million international units, MlU/ml and estradiol less than 40 picogrammes per millilitre (less than 140 picomoles per litre) is confirmatory]. [Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the contraception methods in Section 8.1 if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrollment. For most forms of HRT, at least 2-4 weeks will elapse between the cessation of therapy and the blood draw; this interval depends on the type and dosage of HRT. Following confirmation of their post-menopausal status, they can resume use of HRT during the study without use of a contraceptive method.]
4. Male subjects must agree to use one of the contraception methods listed in Section 8.1. This criterion must be followed from the time of the first dose of study medication until 5 terminal half-lives post-last dose.
5. Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.

6.12 lead ECG without any clinically significant abnormality as judged by the Investigator, and QTc intervals corrected for Bazett ror Fredericia (QTcB and QTcF) less than450 milliseconds (msec)

7.Body weight greater than or equal to 50 kilogrammes (kg) (110 pounds, lbs) for men and greater than or equal to 45 kg (99 lbs) for women and Body Mass Index, BMI within the range 18-30 kilogrammes per squared metre (kg/m2) inclusive.

8.Non-smokers only- Negative urine cotinine test at screening, no history of smoking within 6 months of the start of the study, and with a total pack year history of less than or equal to 1 pack years.

INCLUSION CRITERIA FOR COHORT 4

A subject will be eligible for inclusion in cohort 4 of this study only if all of the following criteria apply:

1. Healthy as determined by the Investigator, based on a medical evaluation including medical history, physical examination, laboratory tests, ECG and Holter assessment at screening. A subject with a clinical abnormality or laboratory parameter outside the reference range for the population being studied may be included only if the Investigator and the GSK Medical Monitor agree that the finding is unlikely to introduce additional risk factors and will not interfere with the study objectives. A subject with a well controlled or mild medical condition (eg controlled hypertension, hypothyroidism adequately treated with replacement therapy, mild chronic obstructive pulmonary disease (COPD) requiring short acting bronchodilators only) may be included only if the Investigator and the GSK Medical Monitor agree that the condition is unlikely to introduce additional risk factors and will not interfere with the study objectives.
2. Male or female (of non child-bearing potential) over 65 years of age inclusive, at the time of signing the informed consent.

   A female subject is eligible to participate only if she is of:

   •Non-childbearing potential defined as pre-menopausal females with a documented tubal ligation (in which case the male partner should use an acceptable form of contraception as specified in section 8.1) or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) > 40 million international units, MlU/ml and estradiol less than 40 picogrammes per millilitre (less than 140 picomoles per litre) is confirmatory]. [Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the contraception methods in Section 8.1 if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrollment. For most forms of HRT, at least 2-4 weeks will elapse between the cessation of therapy and the blood draw; this interval depends on the type and dosage of HRT. Following confirmation of their post-menopausal status, they can resume use of HRT during the study without use of a contraceptive method.]
3. Male subjects must agree to use one of the contraception methods listed in Section 8.1. This criterion must be followed from the time of the first dose of study medication until 5 terminal half-lives post-last dose.
4. Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.

5.12 lead ECG without any clinically significant abnormality as judged by the Investigator and QTcB and QTcF less than 450 msec

6.Body weight greater than or equal to 50 kg (110 lbs) for men and greater than or equal to 45 kg (99lbs) for women and BMI within the range 18-35 kg/m2 inclusive.

7.For non-smokers only - negative urine cotinine test at screening, no history of smoking within 6 months of the start of the study, and with a total pack year history of less than or equal to 1 pack years.

8.For smokers only - a smoking history of greater than or equal to 5 pack years and currently smoking at least 5 cigarettes/day for the last 6 months

EXCLUSION CRITERIA

A subject will not be eligible for inclusion in this study if any of the following criteria apply:

1. A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening
2. Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
3. Significant cardiac, pulmonary, metabolic, renal, gastrointestinal or other conditions that in the opinion of the investigator and/or GSK medical monitor, places the subject at an unacceptable risk as participant in this trial.
4. A positive pre-study drug/alcohol screen.
5. A positive test for human immunodeficiency virus (HIV) antibody.
6. History of regular alcohol consumption within 6 months of the study defined as an average weekly intake of greater than 21 units for males or less than14 units for females. One unit is equivalent to 8 g of alcohol: a half-pint (~240 ml) of beer, 1 glass (125 ml) of wine or 1 (25 ml) measure of spirits.
7. The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 3 months or 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
8. Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
9. Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
10. History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
11. Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
12. Pregnant females as determined by positive serum or urine human Chorionic Gonadotrophin (hCG) test at screening or prior to dosing.
13. Lactating females.
14. Unwillingness or inability to follow the procedures outlined in the protocol.
15. Subject is mentally or legally incapacitated.
16. Consumption of red wine, seville oranges, grapefruit or grapefruit juice and/or pummelos, exotic citrus fruits, grapefruit hybrids or fruit juices from 7 days prior to the first dose of study medication.
17. For non-smokers only - urinary cotinine levels indicative of smoking or history or regular use of tobacco- or nicotine-containing products within 6 months prior to screening.
18. Blood pressure persistently greater than 150 over 90 (150/90) millimetres of mercury (mmHg) at screening.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2009-04-20 (Actual); Primary Completion 2010-06-08 (Actual); Study Completion 2010-06-08 (Actual)

PRIMARY OUTCOMES:
Composite of plasma pharmacokinetic (PK) parameters of GSK2190915 in Cohort 1, 2 and 3 | PK samples will be collected at pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 48 and 72 hours post dose in each period up to 36 days
  PK parameters including area under the plasma concentration-time curve from time zero (pre-dose) extrapolated to infinite time (AUC [0-∞]), Area under the concentration-time curve from time zero (pre-dose) to last time of quantifiable concentration within a subject across all treatments (AUC[0-t]), concentrations at 24h post dose (C24), maximum plasma concentration (Cmax), time to maximum plasma concentration (Tmax), terminal half-life (t1/2) and oral clearance (CL/F) for Cohort 1, 2, 3 will be measured.
Composite of PK parameters in Cohort 4 | Up to 12 days
  PK parameters including area under the plasma concentration-time curve over the dosing interval (AUC [0-tau]), trough C24, Cmax, Tmax, and accumulation for Cohort 4 will be measured.
Composite of PK parameters in Cohort 5 and 6 | PK samples will be collected at pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, and 72 hours post dose in each period up to 36 days
  PK parameters including AUC (0-∞), AUC (0-t), C24, Cmax, Tmax, t1/2 and CL/F for Cohort 5 and 6 will be measured.

SECONDARY OUTCOMES:
Blood pressure measurement for Cohorts 1, 2, and 3 after GSK2190915 administration | Up to 36 days
Blood pressure measurement for Cohorts 4 after GSK2190915 administration | Up to 12 days
Blood pressure measurement for Cohorts 5 and 6 after GSK2190915 administration | Up to 36 days
Pulse rate measurement for Cohorts 1, 2, and 3 after GSK2190915 administration | Up to 36 days
Pulse rate measurement for Cohort 4 after GSK2190915 administration | Up to 12 days
Pulse rate measurement for Cohorts 5 and 6 after GSK2190915 administration | Up to 36 days
ECG measurement for Cohorts 1, 2, 3 after GSK2190915 administration | Up to 36 days
ECG measurement for Cohort 4 after GSK2190915 administration | Up to 12 days
ECG measurement for Cohort 5 and 6 after GSK2190915 administration | Up to 36 days
Holter monitoring for Cohort 4 only after GSK2190915 administration | Up to 12 days
Laboratory assessment for Cohorts 1, 2, 3 after GSK2190915 administration | Up to 36 days
  Laboratory parameters including hematology, clinical chemistry, and urinalysis
Laboratory assessment for Cohort 4 after GSK2190915 administration | Up to 12 days
  Laboratory parameters including hematology, clinical chemistry, and urinalysis
Laboratory assessment for Cohort 5 and 6 after GSK2190915 administration | Up to 36 days
  Laboratory parameters including hematology, clinical chemistry, and urinalysis
Adverse Event reporting for Cohorts 1, 2, and 3 after GSK2190915 administration | Up to 36 days
Adverse Event reporting for Cohort 4 after GSK2190915 administration | Up to 12 days
Adverse Event reporting for Cohorts 5 and 6 after GSK2190915 administration | Up to 36 days

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Results for study 112071 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/112071?search=study&study_ids=112071#rs
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Clinical Study Report: 112071 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 112071 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 112071 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 112071 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 112071 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 112071 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 112071 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register